CLINICAL TRIAL: NCT04751422
Title: A Single-Center Retrospective Study Evaluating Radiofrequency Ablation and Cement Augmentation for the Treatment of Secondary Metastases to the Spine
Brief Title: Medical Data Collection for the Evaluation of Radiofrequency Ablation and Cement Augmentation for the Treatment of Secondary Metastases to the Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1012; NCI-2021-00607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1012 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Malignant Neoplasm in the Spine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (data collection): Patients' medical data is collected retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Medical data is collected

SUMMARY:
This study collects data on the use of radiofrequency ablation and cement augmentation for the treatment of cancer that has spread to the spine (metastases to the spine). Radiofrequency ablation with cement augmentation is a useful approach for the treatment of secondary metastasis to the spine. Information collected in this study may help doctors to learn the effectiveness of this therapy, and may help to evaluate optimal technique, appropriate patient selection, and management of complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the use of radiofrequency ablation and cement augmentation for the treatment of secondary metastases to the spine.

OUTLINE:

Patients' medical data is collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent radiofrequency ablation with cement augmentation at the Department of Interventional Radiology at MD Anderson Cancer Center (MDACC) between 1/1/2017 and 9/26/2020

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent radiofrequency ablation with cement augmentation at the Department of Interventional Radiology at MD Anderson Cancer Center (MDACC) between 1/1/2017 and 9/26/2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | Up to 3 years
  Results will be compared with data available from other published literature.
Clinical success | Up to 3 years
  Results will be compared with data available from other published literature.
Complication rates | Up to 3 years
  Results will be compared with data available from other published literature.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul A Sheth, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org